CLINICAL TRIAL: NCT01046305
Title: Symptom Burden of Patients With Chronic Myeloid Leukemia (CML)
Brief Title: Symptom Burden in Chronic Myeloid Leukemia (CML)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008-0728
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Leukemia
Keywords: Chronic Myeloid Leukemia; CML; Symptom Burden; M. D. Anderson Symptom Inventory; MDASI-CML; Severity; Interference; Questionnaire; Interview
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Part 1: Interview & Questionnaires: Patients interviews and questionnaires about CML symptoms once.
  Interventions: Behavioral: Interview & Questionnaires
- Part 2: Symptoms Rating: Importance of symptoms to CML patients rated by physicians, nurses, patients, and caregivers.
  Interventions: Behavioral: Rating Questionnaire
- Part 3: MDASI-CML Questionnaires: Patients questionnaires about CML symptoms over 1 year using M. D. Anderson Symptom Inventory (MDASI) module (the MDASI-CML)
  Interventions: Behavioral: MDASI-CML Questionnaire

INTERVENTIONS:
Behavioral: Interview & Questionnaires — 30 Minute Interview about what it is like to have CML, followed by symptom questionnaire, quality-of-life questionnaire, and demographic questions taking another 10 minutes for all 3 questionnaires.
  Other Names: Survey
  Groups: Part 1: Interview & Questionnaires
Behavioral: Rating Questionnaire — Questionnaire developed in Part 1 to rate the relevance of symptom items, given to 3-5 physicians, 3-5 nurses, 2-4 patients and their family caregivers, taking about 10 minutes.
  Other Names: Survey; MDASI-CML
  Groups: Part 2: Symptoms Rating
Behavioral: MDASI-CML Questionnaire — Patient questionnaires about CML symptoms over 1 year, completed in person or using Interactive Voice Response (IVR) system every 2 weeks.
  Other Names: Survey; M. D. Anderson Symptom Inventory; MDASI; MDASI-CML
  Groups: Part 3: MDASI-CML Questionnaires

SUMMARY:
Objectives:

The objective of this study is to measure and delineate the symptom burden experienced by patients with chronic myeloid leukemia (CML).

The Primary Aim is to develop and validate an M. D. Anderson Symptom Inventory (MDASI) module (the MDASI-CML), compliant with FDA standards for patient-reported outcomes (PROs), to measure the severity of multiple symptoms and the impact of these symptoms on daily functioning in patients with CML.

The Secondary Aims are:

1. to develop a detailed description of the severity and interference with daily activities of symptoms experienced by patients with CML;
2. to assess the impact of symptom severity in CML on standard functioning and quality of life (QOL) measures including Eastern Cooperative Oncology Group (ECOG) Performance Status and single-item QOL scale;
3. to evaluate the MDASI-CML as an estimate of functional status and QOL in patients with CML;
4. to identify common clusters of symptoms and symptom patterns occurring over multiple measurement time points in patients with CML;

5, to define the qualitative symptom burden of patients with CML;

6. to explore the feasibility of the Interactive Voice Response (IVR) system in measuring symptom severity and interference with daily activities over time in patients with CML.

DETAILED DESCRIPTION:
Part 1:

Interview:

If you agree to take part in this study, while you are at the clinic for a visit, you will be interviewed about what it is like to have CML. The interview should take about 30 minutes to complete.

Questionnaires:

After the interview, you will be asked to answer a symptom questionnaire, a quality-of-life questionnaire, and some demographic questions such as your age and marital status. It will take about 10 minutes to complete all 3 questionnaires.

Length of Study:

After you have completed the interview and questionnaires, your participation on this study will be over.

Additional Information:

The interview will be digitally recorded. The electronic record of the interview will not have your name linked to it and it will be kept on a secure server at M. D. Anderson Cancer Center that is password protected. All study materials will be destroyed after data analysis is completed and study results reported.

Information about your symptoms collected in this study is collected for research purposes only. If you are experiencing severe or troublesome symptoms, you should report them to your doctor or nurse as well as rating them on the symptom assessment questionnaire. If the data collector notices that you have rated a symptom as severe, the data collector will ask you if your doctor or nurse is aware of the symptom or if you intend to report the symptom to your doctor or nurse. If you have not or do not intend to report the symptom, the data collector will let you know that he or she will report the symptom to your doctor or nurse.

This is an investigational study.

Up to 218 participants will take part in this study. Up to 40 will be enrolled in Part 1 of this study. All will be enrolled at MD Anderson.

Part 3:

Symptom Questionnaires:

If you agree to take part in this study, you will complete a questionnaire about any symptoms you are having every 2 weeks for 1 year. On the questionnaire, you will be asked to rate the level of discomfort caused by the symptoms you are having and how the symptoms effect the activities of your daily life. The symptom questionnaire should take about 5 minutes to complete. You will complete the questionnaire during the first study visit and at your clinic visits every 3 months. In between visits, you will be called every 2 weeks to complete the questionnaire by an automated telephone system.

You will decide a convenient time and place for the automated phone system to call you. If you are not available when the automated system calls, it will call you again at a later time. You may also call the automated system if you miss a call. If you are not reached by the automated phone system after several tries, the study staff will call you.

You will be given a secure user name and identification number to use with the automated phone system. You will be shown how the automated phone system works by the study staff.

Two (2) days after the first visit, you will fill out the symptom questionnaire again. You will take it home with you from the clinic with a pre-addressed, stamped envelope given to you by the research staff so you can return it. The research staff will also ask for your telephone number so that they may contact you and remind you to complete the questionnaire.

Quality-of-Life/Demographic Questionnaires:

At the first visit and the 3-month clinic visits, you will also rate your overall quality-of-life. This should take about 1 minute to complete.

At the first visit, you will also be asked some demographic questions (such as your age and marital status). Answering these questions should take about 1 minute.

Opinion Questionnaire:

If you are 1 of the first 30 patients enrolled in the study, at the first visit you will also complete a questionnaire about your opinion of the symptom questionnaire. For example, you will be asked if the symptom questionnaire was easy to understand and to complete and if there were any other questions that should be included. The study staff will use your opinion to decide if other important symptom questions are missing from the questionnaire. This questionnaire should take about 5 minutes to complete.

Length of Study:

You will be on study for 1 year.

Additional Information:

The questionnaires will only use your study number and will not have your name linked to them. All questionnaires and study data will be kept in a locked cabinet at all times. All study materials will be destroyed after data analysis is completed and study results reported.

Information about your symptoms collected in this study is collected for research purposes only. If you are experiencing severe or troublesome symptoms, you should report them to your doctor or nurse as well as rating them on the symptom assessment questionnaire. If the data collector notices that you have rated a symptom as severe, the data collector will ask you if your doctor or nurse is aware of the symptom or if you intend to report the symptom to your doctor or nurse. If you have not or do not intend to report the symptom, the data collector will let you know that he or she will report the symptom to your doctor or nurse.

This is an investigational study.

Up to 218 participants will take part in this study. Up to 160 participants will be enrolled in Part 3 of this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older (Patient and family caregiver only)
2. Ability to speak and read English (All participants)
3. Live in the United States (Patient Phase 3 only)
4. Diagnosis of Philadelphia chromosome positive CML confirmed by pathological and cytogenetic analysis (Patient only)
5. Being followed at M.D. Anderson Cancer Center (Patient only)
6. Consent to participate (All participants)
7. Treatment for CML for at least 1 year (Patient Phase 2 only)
8. Family caregiver also willing to receive packet for expert panel participation (Patient Phase 2 only)
9. Physician or nurse with at least 5 years experience caring for patients with CML (Professional expert only)
10. At least one publication in the last 5 years dealing with CML (Physician professional expert only)
11. Identification as a family caregiver by a patient with CML (Family caregiver only)
12. Patient also willing to receive packet for expert panel participation (Family caregiver only)

Exclusion Criteria:

1. Medical condition or impaired performance status that would preclude participation in the study (Patient only)
2. Diagnosis of active psychosis or severe cognitive impairment as determined by primary physician (Patient only)
3. Active treatment (systemic drug therapy or radiation therapy) for a second malignancy (Patient only Phase 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic myeloid leukemia (CML) patients and their caregivers, 18 years of age or older, physicians and nurses.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Symptom Burden Experienced by CML Patients | Patients followed over 1 year with MDASI-CML questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Loretta A. Williams, PHD, MSN, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Williams LA, Garcia Gonzalez AG, Ault P, Mendoza TR, Sailors ML, Williams JL, Huang F, Nazha A, Kantarjian HM, Cleeland CS, Cortes JE. Measuring the symptom burden associated with the treatment of chronic myeloid leukemia. Blood. 2013 Aug 1;122(5):641-7. doi: 10.1182/blood-2013-01-477687. Epub 2013 Jun 18. PMID 23777764
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org